CLINICAL TRIAL: NCT07069439
Title: Validation and Reliability of the Turkish Version of the Parent-Reported Drug Hypersensitivity Quality of Life Questionnaire (P-DrHy-Q)
Brief Title: Turkish Version of the Parent-Reported Drug Hypersensitivity Quality of Life Questionnaire
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Hilal Gungor, Medical Doctor, Pediatric Immunology and Allergy, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 2025-300613
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-07

CONDITIONS: Drug Hypersensitivity; Quality of Life (QOL); Caregivers; Allergy and Immunology
MeSH Terms: conditions — Drug Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregiver Cohort: This cohort will consist of adult caregivers (parents or legal guardians) of children under 18 years of age with a documented history of drug hypersensitivity. Participants will complete the Turkish version of the Parent-reported Drug Hypersensitivity Quality of Life Questionnaire (P-DrHy-Q) to evaluate its psychometric properties, including internal consistency and test-retest reliability.
  Interventions: Behavioral: Turkish Version of the P-DrHy-Q

INTERVENTIONS:
Behavioral: Turkish Version of the P-DrHy-Q — Participants will complete the Turkish-translated version of the Parent-reported Drug Hypersensitivity Quality of Life Questionnaire (P-DrHy-Q), which includes 12 items assessing psychosocial burden in two domains: mental health and social activity. A subgroup of participants (n ≈ 20) will complete the same questionnaire again after 14 days to assess test-retest reliability

SUMMARY:
This study aims to evaluate the psychometric properties of the Turkish version of the Parent-reported Drug Hypersensitivity Quality of Life Questionnaire (P-DrHy-Q), a disease-specific instrument assessing the health-related quality of life (HRQoL) in caregivers of children with suspected or confirmed drug hypersensitivity reactions. The P-DrHy-Q is designed to capture the psychosocial burden experienced by caregivers and includes two main domains: Mental Health and Social Activity. This study involves a forward-backward translation process, cultural adaptation, internal consistency analysis, and test-retest reliability assessment in a Turkish caregiver population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary caregiver of a child under the age of 18
* Child must have a documented history of drug hypersensitivity
* Fluent in written and spoken Turkish
* Willingness to participate and provide written informed consent
* Availability to complete both baseline and follow-up questionnaire within the designated time frame

Exclusion Criteria:

* Caregivers with diagnosed psychiatric or cognitive disorders
* Inability to read or write in Turkish
* Child currently experiencing an acute drug hypersensitivity reaction
* Previous participation in the pilot testing phase of this validation study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult caregivers (parents or legal guardians) of children under the age of 18 who have a medically confirmed history of drug hypersensitivity. Participants will be recruited from a tertiary care pediatric allergy outpatient clinic. All participants must be fluent in Turkish and able to provide informed consent. The population represents a real-world sample of caregivers managing children with various types of drug allergies, including but not limited to reactions to antibiotics, antipyretics, and nonsteroidal anti-inflammatory drugs (NSAIDs). A subgroup of caregivers will be invited to complete the questionnaire twice to assess test-retest reliability.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Internal Consistency of the Turkish Version of the P-DrHy-Q | Within 30 days from initial questionnaire administration
  The internal consistency of the Turkish translation of the Parent-reported Drug Hypersensitivity Quality of Life Questionnaire (P-DrHy-Q) will be assessed. This analysis will evaluate the degree to which all items on the scale measure the same underlying construct (psychosocial burden in caregivers of children with drug hypersensitivity). Cronbach's alpha coefficient will be calculated for the total scale and its subscales (mental health and social activity).α ≥ 0.70 = Acceptable
Test-Retest Reliability of the Turkish P-DrHy-Q | From Day 1 to Day 15 (14-day interval between two administrations)
  This outcome assesses the stability of the Turkish version of the P-DrHy-Q over time in the absence of clinical change. Test-retest reliability ensures that the questionnaire produces consistent results when administered under similar conditions.A subset of 20 caregivers will complete the P-DrHy-Q a second time after 3 days. The Pearson correlation coefficient will be used to compare scores from the first and second administrations.r ≥ 0.70 = Good-Acceptable

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data (IPD) due to the sensitive nature of patient and caregiver health information. All data will be analyzed and reported in aggregate form to protect participant confidentiality. Only authorized members of the research team will have access to the raw data, which will be stored securely in accordance with institutional and ethical guidelines.